CLINICAL TRIAL: NCT04209855
Title: MIRASOL: A Randomized, Open-label, Phase 3 Study of Mirvetuximab Soravtansine vs. Investigator's Choice of Chemotherapy in Platinum-Resistant, Advanced High-Grade Epithelial Ovarian, Primary Peritoneal, or Fallopian Tube Cancers With High Folate Receptor-Alpha Expression
Brief Title: A Study of Mirvetuximab Soravtansine vs. Investigator's Choice (IC) of Chemotherapy in Platinum-Resistant, Advanced High-Grade Epithelial Ovarian, Primary Peritoneal, or Fallopian Tube Cancers With High Folate Receptor-Alpha (FRα) Expression
Acronym: MIRASOL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: Gynecologic Oncology Group (Network); European Network of Gynaecological Oncological Trial Groups (ENGOT) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMGN853-0416; 2019-003509-80 (EudraCT Number)
Record Dates: First submitted 2019-12-17; First posted 2019-12-24 (Actual); Results first posted 2024-08-01 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Epithelial Ovarian Cancer; Peritoneal Cancer; Fallopian Tube Cancer
Keywords: Platinum-resistant; Folate-receptor alpha expression; Phase 3; Antibody-drug conjugate; mirvetuximab soravtansine; IMGN853; Epithelial Ovarian Cancer; Peritoneal Cancer; Fallopian Tube Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms | interventions — mirvetuximab soravtansine; Paclitaxel; Topotecan; liposomal doxorubicin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Mirvetuximab Soravtansine (Experimental): Participants will receive single-agent mirvetuximab soravtansine (MIRV) at 6 milligrams (mg)/kilogram (kg) adjusted ideal body weight (AIBW) administered intravenously (IV) on Day 1 of every 3-week cycle (Q3W).
  Interventions: Drug: Mirvetuximab Soravtansine
- Investigator's Choice (IC) Chemotherapy (Active Comparator): Participants will receive a dose of IC chemotherapeutic agent calculated using body surface area (BSA). Paclitaxel administered at 80 milligrams/square meter (mg/m^2) as a 1-hour IV infusion on Days 1, 8, 15, and 22 of a 4-week cycle; or topotecan administered at 4 mg/m^2 over 30 minutes on Days 1, 8, and 15 of a 4-week cycle. Alternatively, topotecan could be administered at 1.25 mg/m^2 over 30 minutes on Days 1 to 5 of a 3-week cycle; or pegylated liposomal doxorubicin administered at 40 mg/m^2 as a 1 mg/minute IV infusion on Day 1 of a 4-week cycle. After Cycle 1, if tolerated, pegylated liposomal doxorubicin could be administered as a 1-hour infusion.
  Interventions: Drug: Paclitaxel; Drug: Topotecan; Drug: Pegylated liposomal doxorubicin

INTERVENTIONS:
Drug: Mirvetuximab Soravtansine — Mirvetuximab Soravtansine will be administered per dose and schedule specified in the arm.
  Other Names: MIRV; IMGN853
  Arms: Mirvetuximab Soravtansine
Drug: Paclitaxel — Paclitaxel will be administered per dose and schedule specified in the arm.
  Arms: Investigator's Choice (IC) Chemotherapy
Drug: Topotecan — Topotecan will be administered per dose and schedule specified in the arm.
  Arms: Investigator's Choice (IC) Chemotherapy
Drug: Pegylated liposomal doxorubicin — Pegylated liposomal doxorubicin will be administered per dose and schedule specified in the arm.
  Arms: Investigator's Choice (IC) Chemotherapy

SUMMARY:
This Phase 3 study is designed to compare the efficacy and safety of mirvetuximab soravtansine (MIRV) vs. IC chemotherapy in participants with platinum-resistant high-grade epithelial ovarian cancer, primary peritoneal, or fallopian tube cancer, whose tumors express a high-level of FRα. Participants will be, in the opinion of the Investigator, appropriate for single-agent therapy for their next line of therapy. The FRα positivity will be defined by the Ventana FOLR1 (FOLR1-2.1) CDx assay.

DETAILED DESCRIPTION:
Participants will be randomized to either MIRV or IC chemotherapy (paclitaxel, PEGylated liposomal doxorubicin, or topotecan).

ELIGIBILITY:
Inclusion Criteria:

1. Female participants ≥ 18 years of age
2. Participants must have a confirmed diagnosis of high-grade serious epithelial ovarian cancer, primary peritoneal cancer, or fallopian tube cancer
3. Participants must have platinum-resistant disease:

   1. Participants who have only had 1 line of platinum based therapy must have received at least 4 cycles of platinum, must have had a response (CR or PR) and then progressed between >3 months and ≤ 6 months after the date of the last dose of platinum
   2. Participants who have received 2 or 3 lines of platinum therapy must have progressed on or within 6 months after the date of the last dose of platinum Note: Progression should be calculated from the date of the last administered dose of platinum therapy to the date of the radiographic imaging showing progression. Note: Participants who are platinum-refractory during front-line treatment are excluded
4. Participants must have progressed radiographically on or after their most recent line of therapy
5. Participants must be willing to provide an archival tumor tissue block or slides, or undergo procedure to obtain a new biopsy using a low risk, medically routine procedure for immunohistochemistry (IHC) confirmation of FRα positivity
6. Participant's tumor must be positive for FRα expression as defined by the Ventana FOLR1 (FOLR-2.1) CDx assay
7. Participants must have at least one lesion that meets the definition of measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 (radiologically measured by the Investigator)
8. Participants must have received at least 1 but no more than 3 prior systemic lines of anticancer therapy, and for whom single-agent therapy is appropriate as the next line of treatment:

   1. Adjuvant ± neoadjuvant considered one line of therapy
   2. Maintenance therapy (for example, bevacizumab, poly (ADP-ribose) polymerase [PARP] inhibitors) will be considered as part of the preceding line of therapy (that is, not counted independently)
   3. Therapy changed due to toxicity in the absence of progression will be considered as part of the same line (that is, not counted independently)
   4. Hormonal therapy will be counted as a separate line of therapy unless it was given as maintenance
9. Participant must have an Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 or 1
10. Time from prior therapy:

    1. Systemic antineoplastic therapy (5 half-lives or 4 weeks, whichever is shorter)
    2. Focal radiation completed at least 2 weeks prior to first dose of study drug
11. Participants must have stabilized or recovered (Grade 1 or baseline) from all prior therapy-related toxicities
12. Major surgery must be completed at least 4 weeks prior to first dose and have recovered or stabilized from the side effects of prior surgery
13. Participants must have adequate hematologic, liver and kidney functions defined as:

    1. Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/liter (L) (1,500/microliter [μL]) without granulocyte colony-stimulating factor (G-CSF) in the prior 10 days or long-acting white blood cell (WBC) growth factors in the prior 20 days
    2. Platelet count ≥ 100 x 10^9/L (100,000/μL) without platelet transfusion in the prior 10 days
    3. Hemoglobin ≥ 9.0 g/dL without packed red blood cell (PRBC) transfusion in the prior 21 days
    4. Serum creatinine ≤ 1.5 x upper limit of normal (ULN)
    5. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3.0 x ULN
    6. Serum bilirubin ≤ 1.5 x ULN (participants with documented diagnosis of Gilbert syndrome are eligible if total bilirubin < 3.0 x ULN
    7. Serum albumin ≥ 2 grams (g)/deciliter (dL)
14. Participants or their legally authorized representative must be willing and able to sign the informed consent form (ICF) and to adhere to the protocol requirements
15. Women of childbearing potential (WCBP) must agree to use highly effective contraceptive method(s) while on study drug and for at least 3 months after the last dose of MIRV or at least 6 months after the last dose of paclitaxel, pegylated liposomal doxorubicin, or topotecan
16. WCBP must have a negative pregnancy test within 4 days prior to the first dose of study drug

Exclusion Criteria:

1. Participants with endometrioid, clear cell, mucinous, or sarcomatous histology, mixed tumors containing any of the above histologies, or low-grade or borderline ovarian tumor
2. Participants with primary platinum-refractory disease, defined as disease that did not respond to (CR or PR) or has progressed within 3 months of the last dose of first line platinum-containing chemotherapy
3. Participants with prior wide-field radiotherapy (RT) affecting at least 20% of the bone marrow
4. Participants with > Grade 1 peripheral neuropathy per Common Terminology Criteria for Adverse Events (CTCAE) v5.0
5. Participants with active or chronic corneal disorders, history of corneal transplantation, or active ocular conditions requiring ongoing treatment/monitoring such as uncontrolled glaucoma, wet age-related macular degeneration requiring intravitreal injections, active diabetic retinopathy with macular edema, macular degeneration, presence of papilledema, and /or monocular vision
6. Participants with serious concurrent illness or clinically relevant active infection, including, but not limited to the following:

   1. Active hepatitis B or C infection (whether or not on active antiviral therapy)
   2. Human immunodeficiency virus (HIV) infection
   3. Active cytomegalovirus infection
   4. Any other concurrent infectious disease requiring IV antibiotics within 2 weeks before starting study drug Note: Testing at screening is not required for the above infections unless clinically indicated
7. Participants with history of multiple sclerosis or other demyelinating disease and/or Lambert-Eaton syndrome (paraneoplastic syndrome)
8. Participants with clinically significant cardiac disease including, but not limited to, any one of the following:

   1. Myocardial infarction ≤ 6 months prior to first dose
   2. Unstable angina pectoris
   3. Uncontrolled congestive heart failure (New York Heart Association > class II)
   4. Uncontrolled ≥ Grade 3 hypertension (per CTCAE)
   5. Uncontrolled cardiac arrhythmias
9. Participants assigned to PLD stratum only: Left ventricular ejection fraction (LVEF) below the institutional limit of normal as measured by echocardiography (ECHO) or multigated acquisition (MUGA) scan
10. Participants with a history of hemorrhagic or ischemic stroke within six months prior to randomization
11. Participants with a history of cirrhotic liver disease (Child-Pugh Class B or C)
12. Participants with a previous clinical diagnosis of non-infectious interstitial lung disease (ILD), including noninfectious pneumonitis
13. Participants with required use of folate-containing supplements (for example, folate deficiency)
14. Participants with prior hypersensitivity to monoclonal antibodies
15. Women who are pregnant or lactating
16. Participants with prior treatment with MIRV or other FRα-targeting agents
17. Participants with untreated or symptomatic central nervous system (CNS) metastases
18. Participants with a history of other malignancy within 3 years prior to randomization. Note: does not include tumors with a negligible risk for metastasis or death (for example, adequately controlled basal-cell carcinoma or squamous-cell carcinoma of the skin, or carcinoma in situ of the cervix or breast
19. Prior known hypersensitivity reactions to study drugs and/or any of their excipients
20. People who are detained through a court or administrative decision, receiving psychiatric care against their will, adults who are the subject of a legal protection order (under tutorship/curatorship), people who are unable to express their consent, and people who are subject to a legal guardianship order
21. Simultaneous participation in another research study, in countries or localities where this is the health authority guidance

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 453 (Actual)
Dates: Start 2019-12-31 (Actual); Primary Completion 2023-03-06 (Actual); Study Completion 2024-10-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (214):
- United States (78):
  - University of Alabama at Birmingham (UAB) GYN Oncology, Birmingham, Alabama
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Arizona Oncology Associates, PC - HAL - USOR, Phoenix, Arizona
  - Mayo Clinic, Phoenix, Arizona
  - USOR: Arizona Oncology Associates, PC - HOPE, Tucson, Arizona
  - University of Arizona Cancer Center, Tucson, Arizona
  - UCLA - JCCC Dept of OBGYN - Women's Health Clinical Research Unit, Los Angeles, California
  - Hoag Cancer Center, Newport Beach, California
  - University of California San Francisco, San Francisco, California
  - Olive View - UCLA Medical Center, Sylmar, California
  - Kaiser Permanente Oncology Clinical Trials, Vallejo, California
  - USOR: Rocky Mountain Cancer Centers, Lakewood, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Florida Cancer Specialist South Division, Fort Myers, Florida
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Women's Care Florida / Women's Cancer Associates, St. Petersburg, Florida
  - Florida Cancer Specialist North Division, St. Petersburg, Florida
  - Florida Cancer Specialists, Tallahassee, Florida
  - Florida Cancer Specialist East Division, West Palm Beach, Florida
  - Memorial University Medical Center, Savannah, Georgia
  - Hawaii Pacific Health - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Illinois Cancer Specialists, Arlington Heights, Illinois
  - University of Chicago, Chicago, Illinois
  - Dr. Sudarshan K. Sharma, Ltd., Hinsdale, Illinois
  - Community Health Network, Indianapolis, Indiana
  - University of Kansas Cancer Center, Westwood, Kansas
  - St. Elizabeth Healthcare, Edgewood, Kentucky
  - Norton Cancer Institute, Louisville, Kentucky
  - Ochnser Medical Center Jefferson, New Orleans, Louisiana
  - WK Physicians Network/Gynecologic Oncology Associates, Shreveport, Louisiana
  - Holy Cross Hospital, Silver Spring, Maryland
  - USOR: Maryland Oncology Hematology, P.A., Silver Spring, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - University of Massachusetts, Worcester, Massachusetts
  - St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - USOR: Minnesota Oncology Hematology, PA, Woodbury, Minnesota
  - HCA Midwest Kansas City/ Sarah Cannon, Kansas City, Missouri
  - Sletten Cancer Institute, Great Falls, Montana
  - Center of Hope, Reno, Nevada
  - The Valley Hospital, Inc, Ridgewood, New Jersey
  - Holy Name Medical Center, Teaneck, New Jersey
  - Columbia University Medical Center, New York, New York
  - FirstHealth of the Carolinas Outpatient Cancer Center, Pinehurst, North Carolina
  - USOR: OHC - Oncology_Hematology Care Clinical Trials, Inc., Cincinnati, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Columbus NCORP, Columbus, Ohio
  - Zangmeister Cancer Center, Columbus, Ohio
  - Oncology_Hematology Care Clinical Trials, LLC, Fairfield, Ohio
  - The Ohio State University Wexner Medical Center, Hilliard, Ohio
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute, Tulsa, Oklahoma
  - USOR: Willamette Valley Cancer Institute and Research Center, Eugene, Oregon
  - Legacy Gynecologic Oncology, Portland, Oregon
  - USOR: Northwest Cancer Specialists, P.C., Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Magee-Women's Hospital-UPMC, Pittsburgh, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - Tennessee Oncology / Sarah Cannon Research Institute, Nashville, Tennessee
  - USOR: Texas Oncology-South Austin, Austin, Texas
  - USOR: Texas Oncology - Fort Worth Cancer Center, Fort Worth, Texas
  - University of Texas, Memorial Hermann, Houston, Texas
  - USOR: Texas Oncology - McAllen South Second, McAllen, Texas
  - USOR: Texas Oncology - San Antonio, San Antonio, Texas
  - USOR: Texas Oncology, P.A., Sugar Land, Texas
  - USOR: Texas Oncology - The Woodlands, Gynecologic Oncology, The Woodlands, Texas
  - USOR: Texas Oncology - Tyler, Tyler, Texas
  - USOR: Texas Oncology, P.A., Webster, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - USOR: Virginia Cancer Specialists, PC, Gainesville, Virginia
  - Kadlec Clinic Hematology & Oncology, Kennewick, Washington
  - West Virginia University- MBRCC, Morgantown, West Virginia
- Australia (6):
  - Newcastle Private Hospital, New Lambton Heights, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Monash Health, Clayton, Victoria
  - Oncology Clinics Victoria (OCV) - Cabrini Malvern Hospital Location, Malvern, Victoria
  - Royal North Shore Hospital, Saint Leonards
  - Burnside War Memorial Hospital - The Brian Fricker Oncology Centre, Toorak Gardens
- Belgium (5):
  - OLV Ziekenhuis, Aalst
  - AZ Klina, Brasschaat
  - Universitair Ziekenhuis Antwerpen (UZA) - Borstkliniek, Edegem
  - AZ St-Lucas, Ghent
  - UZ Leuven, Leuven
- Bulgaria (4):
  - Complex Oncology Center, Burgas
  - UMHAT Georgi Stranski, Pleven
  - Acibadem City Clinic Tokuda Hospital, Sofia
  - UMHAT "Sv. Ivan Rilski", EAD, Sofia, Sofia
- Canada (8):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - The Ottawa Hospital General Campus, Ottawa, Ontario
  - Sunnybrook Health Sciences Center, Toronto, Ontario
  - Princess Margaret Cancer Centre - University Health Network, Toronto, Ontario
  - Centre Hospitalier de L'Universite de Montreal, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec
- China (15):
  - Anhui Provincial Cancer Hospital, Hefei, Anhui
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Zhongshan Hospital Xiamen University, Xiamen, Fujian
  - Sun Yat-sen University, Cancer Center, Guangzhou, Guangdong
  - Wuhan Union Hospital of China, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin
  - Liaoning Cancer Hospital, Shenyang, Liaoning
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - Peking University First Hospital, Beijing
  - Beijing Cancer Hospital, Beijing
  - Fudan University Shanghai Cancer Center, Shanghai
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin
- Czechia (3):
  - Fakultní nemocnice Ostrava, Ostrava
  - Všeobecná fakultní nemocnice v Praze, Prague
  - KNTB a.s. Zlín, Zlín
- France (15):
  - Institut Claudius Regaud, Toulouse, Cedex 9
  - Centre Oscar Lambret, Lille, Cedex B.P 307
  - Institut de cancérologie de l'ouest, site Angers, Angers, Cedex
  - CHRU Besançon, Besançon
  - Institut Bergonie, Bordeaux
  - Centre Leon Berard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Cochin Hospital, Paris
  - Groupe Hospitalier Diaconesses Croix Saint-Simon, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Armoricain de radiothérapie, imagerie médicale et oncologie, CARIO, Plérin
  - Institut Curie, Saint-Cloud
  - ICO Centre René Gauducheau, Saint-Herblain
  - Institut de cancérologie de Lorraine, Vandoeuvre Les Nancy_ Cedex
  - Gustave Roussy, Villejuif
- Germany (9):
  - Ulm University Hospital Klinik für Frauenheilkunde und Geburtshilfe, Ulm, Baden-Wurttemberg
  - UMG Göttingen Frauenklinik, Göttingen, Lower Saxony
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden, Saxony
  - Universitätsklinikum Bonn, Bonn
  - Städtisches Klinikum Dessau, Zentrum für Klinische Studien, Dessau
  - Klinikum Dortmund gGmbH / Frauenklinik, Dortmund
  - University Hospital Freiburg, Freiburg im Breisgau
  - UKGM Standort Giessen, Giessen
  - Mammazentrum Hamburg am Krankenhaus Jerusalem, Hamburg
- Israel (6):
  - Wolfson Medical Center, Holon
  - Hadassah Ein Kerem Medical center, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center, Rehovot
  - Ziv Medical Center, Safed
- Italy (11):
  - IOV Istituto Oncologico, Padua, PD
  - Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia, Brescia
  - ASST Lecco- Ospedale A.Manzoni, Lecco
  - IRCCS - Istituto Europeo di Oncologia (The European Institute of Oncology) (IEO), Milan
  - INT Pascale, Naples
  - Centro Operativo Studi Clinici S.C.Oncologia Medica, Perugia
  - Oncologia Azienda Osc-IRCCS Reggio Emilia, Reggio Emilia
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome
  - Azienda Ospedaliera Città Della Salute E Della Scienza Di Torino, Torino
  - Ospedale Mauriziano Umberto I, Torino
  - Istituto Oncologico Candiolo, Torino
- Netherlands (4):
  - Amsterdam UMC, Amsterdam
  - Maastricht UMC, Maastricht
  - Radboud University Medical Center, Nijmegen
  - Erasmus Medical Center, Rotterdam
- Poland (5):
  - Medical University of Gdansk, Gdansk
  - Samodzielny publiczny szpital kliniczny nr 1, Lublin
  - Wojewódzki Szpital Specjalistyczny, Oddzial Kliniczny Ginekologii Onkologiczne, Olsztyn
  - Wielkopolskie Centrum Onkologii, Poznan
  - Szpital Kliniczny im. Ks. Anny Mazowieckiej, Warsaw
- Portugal (4):
  - Fundação Champalimaud, Lisbon
  - Hospital da Luz, S.A, Lisbon
  - Centro Hospitalar de Lisboa Norte, E.P.E. - Hospital de Santa Maria, Lisbon
  - Hospital Beatriz Angelo, Loures
- Russia (4):
  - BIH of Omsk Region "Clinical Oncology Dispensary", Omsk, Omsk Oblast
  - LLC "VitaMed", Moscow
  - Leningrad regional oncology dispensa, Saint Petersburg
  - State Autonomous Healthcare Institution Republican Clinical Oncological Dispensary of the MoH of Republic Bashkortostan, Ufa
- Serbia (3):
  - Oncology and Radiology Institute Serbia, Belgrade
  - Oncology Institute Vojvodina, Surgical Oncology Clinic, Kamenitz
  - Clinical Center Kragujevac, Kragujevac
- South Korea (6):
  - National Cancer Center - Center for Uterine Cancer, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - University of Ulsan College of Medicine - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (12):
  - Hospital Clínico de Santiago, Santiago de Compostela, A Coruña
  - H. U. de Jaén, Jaén, Andalusia
  - Hospital Universitario Infanta Sofía, San Sebastián de los Reyes, Madrid
  - Institut Català d'Oncologia, Badalona
  - Hospital Provincial de Castellon, Castelló
  - H. San Pedro de Alcántara, Cáceres
  - Hospital de San Chinarro-Clara Campal, Madrid
  - Hospital Clínico Universitario Virgen de la Arrixaca, Murcia
  - Parc Taulí, Sabadell
  - Virgen del Rocío, Seville
  - Hospital de la Fe, Valencia
  - HCU Lozano Blesa, Zaragoza
- Taiwan (3):
  - Far Eastern Memorial Hospital, New Taipei City
  - Mackay Memorial Hospital - Taipei Branch, Taipei
  - Taipei Veterans General Hospital, Taipei
- Ukraine (5):
  - Chernihiv Medical Center of Modern Oncology of Chernihiv Regional Council, Chernihiv, Chernihiv Oblast
  - Grigoriev Institute for Medical Radiology NAMS of Ukraine, Kharkiv, Kharkivs’ka Oblast’
  - Communal non-profit enterprise "Khmelnytskyi Regional Antitumor Center" of Khmelnytskoyi Regional Council, Khmelnytskyi, Khmelnytskyi Oblast
  - Communal non-profit enterprise "Cherkasy Regional Oncology Dispensary of Cherkasy oblast council", Cherkasy
  - Prykarpatskyi Clinical Oncology Center of Ivano-Frankivsk Regional Council, Ivano-Frankivsk
- United Kingdom (8):
  - Peterborough City Hospital, Peterborough, Cambridgeshire
  - Royal Devon and Exeter Hospital (Wonford), Exeter, Devon
  - University Hospitals Coventry and Warwickshire, Coventry
  - Beatson West of Scotland Cancer Centre, Glasgow
  - St Bartholomew's Hospital-Barts Health NHS Trust, London
  - University College London Hospital, London
  - The Royal Marsden NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester

REFERENCES:
- [Derived] Van Gorp T, Moore KN, Konecny GE, Leary A, Garcia-Garcia Y, Banerjee S, Lorusso D, Lee JY, Moroney JW, Caruso G, Klasa-Mazurkiewicz D, Tromp J, Martin LP, Breuer S, Leath CA 3rd, Cibula D, Weroha SJ, Estevez-Garcia P, O'Malley DM, Miller RE, Coffman L, Scandurra G, Berton D, Li L, Zagadailov E, Diver EJ, Tredan O, Hilpert F. Patient-reported outcomes from the MIRASOL trial evaluating mirvetuximab soravtansine versus chemotherapy in patients with folate receptor alpha-positive, platinum-resistant ovarian cancer: a randomised, open-label, phase 3 trial. Lancet Oncol. 2025 Apr;26(4):503-515. doi: 10.1016/S1470-2045(25)00021-X. PMID 40179908
- [Derived] Moore KN, Angelergues A, Konecny GE, Garcia Y, Banerjee S, Lorusso D, Lee JY, Moroney JW, Colombo N, Roszak A, Tromp J, Myers T, Lee JW, Beiner M, Cosgrove CM, Cibula D, Martin LP, Sabatier R, Buscema J, Estevez-Garcia P, Coffman L, Nicum S, Duska LR, Pignata S, Galvez F, Wang Y, Method M, Berkenblit A, Bello Roufai D, Van Gorp T; Gynecologic Oncology Group Partners and the European Network of Gynaecological Oncological Trial Groups. Mirvetuximab Soravtansine in FRalpha-Positive, Platinum-Resistant Ovarian Cancer. N Engl J Med. 2023 Dec 7;389(23):2162-2174. doi: 10.1056/NEJMoa2309169. PMID 38055253

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 453 participants were randomized to a treatment group and included in the Intent-to-Treat (ITT) population. 425 participants received at least 1 dose of study drug and were included in the Safety Population.
Groups:
- Mirvetuximab Soravtansine: Participants received single-agent mirvetuximab soravtansine (MIRV) at 6 milligrams (mg)/kilogram (kg) adjusted ideal body weight (AIBW) administered intravenously (IV) on Day 1 of every 3-week cycle (Q3W).
- Investigator's Choice (IC) Chemotherapy: Participants received a dose of IC chemotherapeutic agent calculated using body surface area (BSA). Paclitaxel administered at 80 milligrams/square meter (mg/m^2) as a 1-hour IV infusion on Days 1, 8, 15, and 22 of a 4-week cycle; or topotecan administered at 4 mg/m^2 over 30 minutes on Days 1, 8, and 15 of a 4-week cycle. Alternatively, topotecan could have been administered at 1.25 mg/m^2 over 30 minutes on Days 1 to 5 of a 3-week cycle; or pegylated liposomal doxorubicin administered at 40 mg/m^2 as a 1 mg/minute IV infusion on Day 1 of a 4-week cycle. After Cycle 1, if tolerated, pegylated liposomal doxorubicin could have been administered as a 1-hour infusion.
Period: Overall Study
Arm/Group | Mirvetuximab Soravtansine | Investigator's Choice (IC) Chemotherapy
Started | 227 | 226
Received at Least 1 Dose of Study Drug | 218 | 207
Completed (Still on treatment) | 0 | 0
Not Completed | 227 | 226
Not completed — Death | 161 | 177
Not completed — PI Discretion | 1 | 1
Not completed — Lost to Follow-up | 5 | 2
Not completed — Withdrew consent | 10 | 24
Not completed — Sponsor decision | 44 | 18
Not completed — Other than specified | 6 | 4

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population included all participants randomized to the study, regardless of whether or not participants received study treatment (MIRV or IC Chemo).
Groups:
- Mirvetuximab Soravtansine: Participants received single-agent MIRV at 6 mg/kg AIBW administered IV on Day 1 of Q3W.
- Investigator's Choice (IC) Chemotherapy: Participants received a dose of IC chemotherapeutic agent calculated using BSA. Paclitaxel administered at 80 mg/m^2 as a 1-hour IV infusion on Days 1, 8, 15, and 22 of a 4-week cycle; or topotecan administered at 4 mg/m^2 over 30 minutes on Days 1, 8, and 15 of a 4-week cycle. Alternatively, topotecan could have been administered at 1.25 mg/m^2 over 30 minutes on Days 1 to 5 of a 3-week cycle; or pegylated liposomal doxorubicin administered at 40 mg/m^2 as a 1 mg/minute IV infusion on Day 1 of a 4-week cycle. After Cycle 1, if tolerated, pegylated liposomal doxorubicin could have been administered as a 1-hour infusion.
- Total: Total of all reporting groups
Arm/Group | Mirvetuximab Soravtansine | Investigator's Choice (IC) Chemotherapy | Total
Number analyzed (Participants) | 227 | 226 | 453
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.3 (9.85) | 62.3 (9.30) | 62.8 (9.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 227 | 226 | 453
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 15 | 27
  Not Hispanic or Latino | 177 | 163 | 340
  Unknown or Not Reported | 38 | 48 | 86
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 28 | 25 | 53
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 5 | 13
  White | 156 | 145 | 301
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 35 | 51 | 86

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) as Assessed by Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Description: PFS was defined as the time from randomization until progressive disease (PD) or death whichever occurred first. PD: At least a 20% increase in the sum of the longest diameters (SoD) of target lesion, taken as reference the smallest (nadir) SoD since and including baseline. In addition to the relative increase of 20%, the SoD must also demonstrate an absolute increase of at least 5 millimeters (mm). Unequivocal progression of non-target lesions and appearance of new lesions. Unequivocal progression should not normally trump target lesion status. It must be representative of overall disease status change, not a single lesion increase.
Time Frame: From randomization until PD or death, whichever occurred first (up to approximately 36 months)
Population: The ITT population included all participants randomized to the study, regardless of whether or not participants received study treatment (MIRV or IC Chemo).
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Mirvetuximab Soravtansine: Participants randomized to single-agent MIRV at 6 mg/kg AIBW administered IV on Day 1 of Q3W.
- Investigator's Choice (IC) Chemotherapy: Participants randomized to IC chemotherapeutic agent calculated using BSA. Paclitaxel administered at 80 mg/m^2 as a 1-hour IV infusion on Days 1, 8, 15, and 22 of a 4-week cycle; or topotecan administered at 4 mg/m^2 over 30 minutes on Days 1, 8, and 15 of a 4-week cycle. Alternatively, topotecan could have been administered at 1.25 mg/m^2 over 30 minutes on Days 1 to 5 of a 3-week cycle; or pegylated liposomal doxorubicin administered at 40 mg/m^2 as a 1 mg/minute IV infusion on Day 1 of a 4-week cycle. After Cycle 1, if tolerated, pegylated liposomal doxorubicin could have been administered as a 1-hour infusion.
Arm/Group | Mirvetuximab Soravtansine | Investigator's Choice (IC) Chemotherapy
Number analyzed (Participants) | 227 | 226
months | 5.59 [4.34 to 5.88] | 3.98 [2.86 to 4.47]
Statistical Analysis 1: Comparison: Mirvetuximab Soravtansine vs Investigator's Choice (IC) Chemotherapy; Test type: Superiority; p < 0.0001, Log Rank; Cox Proportional Hazard = 0.63, 95% CI 2-sided [0.513 to 0.785]

2. Secondary Outcome: Objective Response Rate (ORR), as Assessed by the Investigator Using RECIST v1.1
Description: ORR was defined as percentage of participants with a confirmed best overall response (BOR) of complete response (CR) or partial response (PR). CR: Disappearance of all target or non-target lesions. All pathological or non-pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR: At least 30% decrease in the sum of the longest diameters (SoD) of target lesions, taking as reference the baseline SoD.
Time Frame: Up to approximately 36 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Mirvetuximab Soravtansine | Investigator's Choice (IC) Chemotherapy
Number analyzed (Participants) | 227 | 226
percentage of participants | 41.9 [35.4 to 48.6] | 15.9 [11.4 to 21.4]

3. Secondary Outcome: Overall Survival Assessed by the Investigator Using RECIST v1.1
Description: Overall survival was defined as the time from the date of first dose until the date of death from any cause, estimated using the Kaplan-Meier method.
Time Frame: Up to approximately 45 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Mirvetuximab Soravtansine | Investigator's Choice (IC) Chemotherapy
Number analyzed (Participants) | 227 | 226
months | 16.85 [14.36 to 19.78] | 13.34 [11.37 to 15.15]

4. Secondary Outcome: Number of Participants Achieving at Least 15 Point Absolute Improvement in the Abdominal/Gastrointestinal (GI) Scale of European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire - Ovarian Cancer Module 28 (QLQ-OV28)
Description: The EORTC QLQ-OV28 is specific for ovarian cancer and consists of 28 items assessing abdominal/gastrointestinal symptoms (6 items), peripheral neuropathy (2 items), other chemotherapy side effects (5 items), hormonal symptoms (2 items), body image (2 items), attitudes to disease/treatment (3 items), sexuality (4 items) and 4 other single items. Each scale was scored from 0 to 100 with higher scores on the symptom scales indicating greater symptom burden. Higher scores represent a higher ("better") level of functioning. Presented here are the number of participants achieving at least 15 point absolute improvement at Week 8 or Week 9 in the abdominal/GI scale of the EORTC QLQ-OV28.
Time Frame: Baseline and Week 8 or 9
Population: The ITT population included all participants randomized to the study, regardless of whether or not participants received study treatment (MIRV or IC Chemo). Here, "Overall Number of Participants Analyzed" is the number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Mirvetuximab Soravtansine | Investigator's Choice (IC) Chemotherapy
Number analyzed (Participants) | 162 | 150
Participants | 34 | 23

5. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence that developed or worsened in severity during the conduct of a clinical study and did not necessarily have a causal relationship to study drug. TEAEs were defined as AEs with an onset date on or after the first dose of study drug, and within 30 days of the last dose of study drug or prior to the start of a new anticancer treatment, whichever occurred first. A summary of serious and all other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Up to approximately 37 months
Population: The Safety Population included all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Mirvetuximab Soravtansine | Investigator's Choice (IC) Chemotherapy
Number analyzed (Participants) | 218 | 207
Participants | 211 | 194

6. Secondary Outcome: Duration of Response (DOR) as Assessed by the Investigator Using RECIST v1.1
Description: DOR was defined as the time from the date of the first response (CR or PR), until the date of PD or death from any cause, whichever occurred first. DOR for participants who have not progressed or died at the time of analysis are censored at the date of their last tumor assessment. PD: At least a 20% increase in the SoD of target lesion, taken as reference the smallest (nadir) SoD since and including baseline. In addition to the relative increase of 20%, the SoD must also have demonstrated an absolute increase of at least 5 mm. DOR was estimated using the Kaplan-Meier method.
Time Frame: Up to approximately 34 months
Population: The ITT population included all participants randomized to the study, regardless of whether or not participants received study treatment (MIRV or IC Chemo). Here, "Overall number of participants analyzed" is the number of evaluable participants for this outcome measure who had CR or PR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Mirvetuximab Soravtansine | Investigator's Choice (IC) Chemotherapy
Number analyzed (Participants) | 95 | 36
months | 6.93 [5.78 to 8.84] | 4.44 [4.17 to 5.75]

7. Secondary Outcome: Percentage of Participants With Cancer Antigen 125 (CA-125) Confirmed Clinical Response Per Gynecologic Cancer Intergroup (GCIG) Criteria
Description: The GCIG CA-125 response was defined as at least 50% reduction in CA-125 levels from baseline. The response must have been confirmed and maintained for at least 28 days.
Time Frame: Baseline up to approximately 36 months
Population: The CA-125-Evaluable Population included all randomized participants who received at least 1 dose of MIRV or IC Chemo, whose pretreatment CA-125 was ≥ 2.0 times the upper limit of normal (ULN), within 2 weeks prior to randomization, and who had at least 1 post-baseline CA-125 evaluation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Mirvetuximab Soravtansine | Investigator's Choice (IC) Chemotherapy
Number analyzed (Participants) | 181 | 156
percentage of participants | 58.0 [50.5 to 65.3] | 30.1 [23.1 to 38.0]

8. Secondary Outcome: Time to Second Progression-Free Survival (PFS 2)
Description: PFS 2 was defined as the time from date of randomization until second disease progression or death whichever occurred first.
Time Frame: Up to approximately 44 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Mirvetuximab Soravtansine | Investigator's Choice (IC) Chemotherapy
Number analyzed (Participants) | 227 | 226
months | 11.01 [9.30 to 12.02] | 7.59 [6.60 to 8.84]

ADVERSE EVENTS:
Time Frame: All-cause mortality and adverse event tables include events reported from the start of safety data collection to the end of the study. The median time on follow-up was 31.1 months and 29.7 months for Mirvetuximab Soravtansine and Investigator's Choice (IC) Chemotherapy, respectively.
Arm/Group | Mirvetuximab Soravtansine | Investigator's Choice (IC) Chemotherapy
All-Cause Mortality (participants affected / at risk) | 162/227 | 177/226
Serious Adverse Events (participants affected / at risk) | 62/227 | 73/226
Other Adverse Events (participants affected / at risk) | 212/227 | 196/226
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mirvetuximab Soravtansine (N=227) | Investigator's Choice (IC) Chemotherapy (N=226)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 4 (6)
PANCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 3 (5) | 3 (3)
CARDIOPULMONARY FAILURE (Cardiac disorders) | 1 (1) | 0 (0)
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 (0) | 1 (1)
CORONARY ARTERY STENOSIS (Cardiac disorders) | 1 (1) | 0 (0)
PERICARDIAL EFFUSION (Cardiac disorders) | 1 (1) | 1 (1)
KERATITIS (Eye disorders) | 1 (1) | 0 (0)
KERATOPATHY (Eye disorders) | 1 (1) | 0 (0)
RETINAL DETACHMENT (Eye disorders) | 1 (1) | 0 (0)
ABDOMINAL HERNIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 6 (6) | 1 (1)
ASCITES (Gastrointestinal disorders) | 4 (5) | 2 (2)
CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 1 (2) | 0 (0)
ENTEROCUTANEOUS FISTULA (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTROINTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 (0) | 1 (1)
HAEMORRHOIDAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
HAEMORRHOIDS (Gastrointestinal disorders) | 1 (1) | 0 (0)
ILEUS (Gastrointestinal disorders) | 1 (1) | 0 (0)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 5 (6) | 6 (7)
LARGE INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 1 (1)
MALIGNANT GASTROINTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 1 (1)
OBSTRUCTION GASTRIC (Gastrointestinal disorders) | 0 (0) | 1 (1)
OESOPHAGITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
PNEUMOPERITONEUM (Gastrointestinal disorders) | 1 (1) | 0 (0)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 6 (7) | 11 (12)
SUBILEUS (Gastrointestinal disorders) | 1 (1) | 3 (5)
VOMITING (Gastrointestinal disorders) | 3 (3) | 2 (2)
ASTHENIA (General disorders) | 3 (3) | 0 (0)
COMPLICATION ASSOCIATED WITH DEVICE (General disorders) | 1 (1) | 0 (0)
DISEASE PROGRESSION (General disorders) | 0 (0) | 1 (1)
FATIGUE (General disorders) | 2 (4) | 2 (5)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 3 (3) | 2 (3)
PYREXIA (General disorders) | 2 (2) | 2 (3)
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 1 (1) | 0 (0)
IMMUNE-MEDIATED ADVERSE REACTION (Immune system disorders) | 1 (1) | 0 (0)
BACTERAEMIA (Infections and infestations) | 0 (0) | 1 (1)
BACTERIAL SEPSIS (Infections and infestations) | 1 (1) | 0 (0)
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 2 (2) | 1 (2)
COVID-19 PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1)
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 2 (2)
GASTROENTERITIS VIRAL (Infections and infestations) | 0 (0) | 1 (1)
KIDNEY INFECTION (Infections and infestations) | 0 (0) | 1 (1)
METAPNEUMOVIRUS PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1)
NEUTROPENIC SEPSIS (Infections and infestations) | 1 (1) | 0 (0)
PERITONITIS (Infections and infestations) | 1 (1) | 1 (1)
PERITONITIS BACTERIAL (Infections and infestations) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 1 (1) | 2 (2)
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 1 (1) | 0 (0)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0)
SEPSIS (Infections and infestations) | 1 (1) | 0 (0)
SEPTIC SHOCK (Infections and infestations) | 0 (0) | 2 (3)
SINUSITIS (Infections and infestations) | 0 (0) | 1 (1)
SUSPECTED COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
HEAD INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
PROCEDURAL PNEUMOTHORAX (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
ULNA FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OXYGEN SATURATION DECREASED (Investigations) | 0 (0) | 1 (1)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 0 (0) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPOVOLAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
MALNUTRITION (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
METASTASES TO CENTRAL NERVOUS SYSTEM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
ONCOLOGIC COMPLICATION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OVARIAN CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
TUMOUR ASSOCIATED FEVER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 (0) | 1 (1)
DIZZINESS (Nervous system disorders) | 1 (1) | 0 (0)
ISCHAEMIC STROKE (Nervous system disorders) | 1 (1) | 0 (0)
PERIPHERAL SENSORIMOTOR NEUROPATHY (Nervous system disorders) | 1 (1) | 0 (0)
RENAL FAILURE (Renal and urinary disorders) | 0 (0) | 1 (1)
URINARY TRACT OBSTRUCTION (Renal and urinary disorders) | 0 (0) | 1 (1)
INTERMENSTRUAL BLEEDING (Reproductive system and breast disorders) | 0 (0) | 1 (1)
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 1 (1) | 0 (0)
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
HYDROTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 1 (1)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1)
HYPERTENSION (Vascular disorders) | 1 (1) | 0 (0)
PERIPHERAL ISCHAEMIA (Vascular disorders) | 1 (1) | 0 (0)
VENA CAVA THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mirvetuximab Soravtansine (N=227) | Investigator's Choice (IC) Chemotherapy (N=226)
ANAEMIA (Blood and lymphatic system disorders) | 30 (66) | 79 (212)
LEUKOPENIA (Blood and lymphatic system disorders) | 3 (3) | 12 (34)
NEUTROPENIA (Blood and lymphatic system disorders) | 27 (49) | 62 (185)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 16 (20) | 35 (81)
CATARACT (Eye disorders) | 67 (132) | 28 (31)
DRY EYE (Eye disorders) | 73 (149) | 15 (17)
EYE PAIN (Eye disorders) | 21 (29) | 1 (2)
KERATOPATHY (Eye disorders) | 78 (211) | 4 (6)
PHOTOPHOBIA (Eye disorders) | 46 (73) | 4 (4)
VISION BLURRED (Eye disorders) | 101 (297) | 12 (14)
VISUAL ACUITY REDUCED (Eye disorders) | 29 (53) | 0 (0)
VITREOUS FLOATERS (Eye disorders) | 17 (23) | 7 (7)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 16 (17) | 12 (15)
ABDOMINAL PAIN (Gastrointestinal disorders) | 65 (102) | 35 (48)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 15 (18) | 12 (15)
CONSTIPATION (Gastrointestinal disorders) | 65 (87) | 44 (66)
DIARRHOEA (Gastrointestinal disorders) | 68 (111) | 37 (62)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 13 (17) | 6 (8)
NAUSEA (Gastrointestinal disorders) | 61 (95) | 63 (93)
STOMATITIS (Gastrointestinal disorders) | 9 (13) | 23 (30)
VOMITING (Gastrointestinal disorders) | 40 (56) | 37 (49)
ASTHENIA (General disorders) | 39 (72) | 38 (60)
FATIGUE (General disorders) | 67 (96) | 51 (94)
OEDEMA PERIPHERAL (General disorders) | 13 (15) | 18 (25)
PYREXIA (General disorders) | 12 (16) | 12 (13)
COVID-19 (Infections and infestations) | 19 (19) | 11 (11)
URINARY TRACT INFECTION (Infections and infestations) | 20 (24) | 21 (27)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 22 (36) | 11 (15)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 25 (46) | 13 (14)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 12 (19) | 6 (10)
BLOOD CREATININE INCREASED (Investigations) | 4 (6) | 12 (20)
WEIGHT DECREASED (Investigations) | 22 (30) | 8 (10)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 7 (15) | 18 (72)
DECREASED APPETITE (Metabolism and nutrition disorders) | 44 (67) | 29 (32)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 16 (23) | 15 (24)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 12 (18) | 19 (24)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 35 (47) | 12 (13)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 25 (29) | 18 (22)
MYALGIA (Musculoskeletal and connective tissue disorders) | 21 (29) | 8 (11)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 15 (20) | 13 (13)
DYSGEUSIA (Nervous system disorders) | 12 (14) | 10 (10)
HEADACHE (Nervous system disorders) | 31 (39) | 20 (25)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 50 (75) | 31 (60)
PARAESTHESIA (Nervous system disorders) | 12 (16) | 1 (1)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 21 (36) | 12 (21)
INSOMNIA (Psychiatric disorders) | 12 (14) | 7 (16)
COUGH (Respiratory, thoracic and mediastinal disorders) | 25 (31) | 18 (22)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 18 (21) | 24 (31)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 19 (23)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 15 (22) | 1 (2)
ALOPECIA (Skin and subcutaneous tissue disorders) | 4 (4) | 30 (35)
DRY SKIN (Skin and subcutaneous tissue disorders) | 3 (3) | 17 (18)
HYPERTENSION (Vascular disorders) | 13 (19) | 8 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2020-12-10): https://cdn.clinicaltrials.gov/large-docs/55/NCT04209855/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-14): https://cdn.clinicaltrials.gov/large-docs/55/NCT04209855/SAP_001.pdf